CLINICAL TRIAL: NCT06572514
Title: The Exploratory Study of the Feasibility of De-escalating Radiation Strategy After NAC in Combination With Immunotherapy in LAHNSCC
Brief Title: De-escalation Radiation Strategy After NAC in Combination With ICI in LAHNSCC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, GAOYUNSHENG, Principal Investigator, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAHNSCC-02
Record Dates: First submitted 2023-12-17; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): Eligible patients received two cycles of pembrolizumab immunotherapy in combination with albumin-bound paclitaxel and cisplatin induction chemotherapy, followed by definitive concurrent radiochemotherapy.
  Interventions: Drug: immunotherapy：pembrolizumab；chemo：albumin-bound paclitaxel and cisplatin

INTERVENTIONS:
Drug: immunotherapy：pembrolizumab；chemo：albumin-bound paclitaxel and cisplatin — The immunotherapy drug was pembrolizumab at a dose of 200 mg, administered on the first day of each cycle every 3 weeks. The induction chemotherapy regimen included albumin-bound paclitaxel at 260 mg/m2 and cisplatin at 75 mg/m2, given every 3 weeks, either concurrently with immunotherapy or on the second day.
  Other Names: definitive radiation

SUMMARY:
This study is a single-arm exploratory study conducted in LAHNSCC. Eligible patients received two cycles of pembrolizumab immunotherapy in combination with albumin-bound paclitaxel and cisplatin induction chemotherapy, followed by definitive concurrent radiochemotherapy. Three months after the completion of radiotherapy, a follow-up examination was conducted, and salvage surgery or systemic therapy was performed as necessary based on the follow-up results.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, with medical decision-making capacity
2. Signed informed consent
3. ECOG score of 0-1
4. Pathologically diagnosed with oral cancer, oropharyngeal cancer, laryngeal cancer, or hypopharyngeal cancer
5. Exclusion of distant metastasis
6. Clearly evaluable lesion (per RECIST 1.1 criteria)
7. Expected life span ≥6 months
8. Laboratory test results meet the following requirements: WBC ≥ 3×10^9/L, ANC ≥ 2.0×10^9/L, PLT ≥ 80×10^9/L, Hb ≥ 80g/L (according to the normal standards of the central laboratory); Liver function: Total bilirubin, ALT, and AST all ≤ 1.5x UNL (upper normal limit); AST (SGOT)/ALT (SGPT) ≤ 2.5 x IULN (upper normal limit); Kidney function: Cr ≤ 1.5x UNL (upper normal limit), and creatinine clearance rate ≥ 60 ml/min (calculated using the Cockcroft and Gault formula); Thyroid function T3 and T4 within the normal range (hypothyroidism can be corrected with oral thyroid hormone supplementation); Heart function: All three cardiac enzymes and pro-BNP within the normal range, no history of heart attack; Adrenal function: Normal cortisol secretion function or correctable based on endocrine assessment
9. HBV-infected patients with HBV-DNA copy numbers less than 500 IU/ml
10. No history of other malignant tumors in the past 5 years (excluding basal cell carcinoma of the skin and thyroid cancer).

Exclusion Criteria:

1. No indications for curative radiotherapy or contraindications to radiochemotherapy.
2. Clinical factors identified by the investigator that could potentially affect the completion of the study protocol (such as bleeding, active infection, or mental factors).
3. Patients requiring long-term maintenance steroid therapy (including oral and intravenous use); local use or inhalation can be included in the study.
4. Previous history of autoimmune diseases or in the active phase of the disease [including but not limited to inflammatory bowel disease (IBD), rheumatoid arthritis, autoimmune hepatitis, systemic sclerosis (scleroderma and its variants), systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathies (such as Guillain-Barré syndrome)], vitiligo, and correctable endocrine deficiencies such as hypothyroidism and physiological cortisol deficiency can be included in the study and are not exclusion criteria.
5. History of active tuberculosis or non-infectious pneumonia or any clinical evidence.
6. Active phase of viral hepatitis, HBV DNA > 500 IU/ml.
7. Acquired Immunodeficiency Syndrome (AIDS).
8. Concurrent severe medical conditions (including heart diseases) with coexisting diseases or conditions affecting the patient's normal enrollment or safety during the study.
9. Prior immunotherapy for other tumors.
10. History of other malignant tumors within 5 years (excluding cured basal cell carcinoma of the skin or thyroid cancer).
11. Pregnant or lactating women.
12. Concurrently suffering from other malignant tumors.
13. Cannot or unwilling to sign the informed consent form.
14. Vaccination within 4 weeks.
15. Allergic reaction to the investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 1 year
  Progression-free survival (PFS) (local-regional recurrence) is defined as the time from enrollment to the occurrence of local or regional lymph node recurrence or death for any reason.

SECONDARY OUTCOMES:
Overall survival (OS) | 3-year
  Overall survival is defined as the time from enrollment to death for any reason
Clinical response rate | 6 months
  Clinical response is defined as the radiological evaluation of tumor regression as partial remission (PR) and complete remission (CR) on imaging assessment three months after the completion of treatment.
Safety(Grade 3-5 AE) | 1-year
  Safety is primarily assessed based on the probability of occurrence of Grade 3-5 adverse effects in different organs according to CTCAE 4.0 (including radiation-related injuries and adverse reactions to immunotherapy).
Quality of life | 6 month and 1 year after the treatment
  The assessment of quality of life is conducted using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Head and Neck Module (EORTC QLQ-H&N 35), which includes eight domains: pain, swallowing, senses, speech, social eating, social contact, sexuality and single items. Each item is scored on a scale from 0 to 100. A high score for a functional scale or global QOL implies a high level of functioning or global QOL, whereas a high score for a symptom scale or single item implies a high level of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No